CLINICAL TRIAL: NCT04075266
Title: An Open-Label, Parallel-Group Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of Ocrelizumab in Children and Adolescents With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study of Ocrelizumab in Children and Adolescents With Relapsing-Remitting Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA39085; 2016-002667-34 (EudraCT Number)
Record Dates: First submitted 2019-08-14; First posted 2019-08-30 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants with a body weight from >/= 25 kg to < 40 kg (with at least 2 participants with a body weight from >/= 25 kg to </= 35 kg) will receive 300 milligram (mg) ocrelizumab
  Interventions: Drug: Ocrelizumab
- Cohort 2 (Experimental): Participants with a body weight >/= 40 kg (with at least 2 participants with a body weight >/= 40 kg but </= 50 kg) will receive 600 mg ocrelizumab
  Interventions: Drug: Ocrelizumab
- Cohort 3 (optional) (Experimental): Based on PK, PD, safety, and tolerability data analyses of Cohorts 1 and 2, additional participants with a body weight from >/= 25 kg to < 40 kg may be enrolled and receive another dose level of ocrelizumab
  Interventions: Drug: Ocrelizumab
- Cohort 4 (optional) (Experimental): Based on PK, PD, safety, and tolerability data analyses of Cohorts 1 and 2, additional participants with a body weight >/= 40 kg may be enrolled and receive another dose level of ocrelizumab
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab is administered as two infusions of half the dose given 14 days apart for the first dose, then subsequent doses are administered as a single infusion every 24 weeks.
  Cohort 1: total dose of 300 mg Cohort 2: total dose of 600 mg Cohort 3 and 4: additional dose level(s) may be lower than 300 mg, between 300 mg and 600 mg, or higher than 600 mg, but will be no higher than 1200 mg

SUMMARY:
This 2-year study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic (PD) effects of ocrelizumab in children and adolescents ages ≥ 10 to ≤ 18 years with relapsing-remitting multiple sclerosis (RRMS). The data from this study will serve to determine the dosing regimen of ocrelizumab to be further investigated in the subsequent Phase III study in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >/= 25 kg
* Children and adolescents must have received all childhood required vaccinations
* Female participants of childbearing potential must agree to either remain completely abstinent or to use reliable means of contraception
* Diagnosis of relapsing-remitting multiple sclerosis (RRMS)
* Expanded Disability Status Scale (EDSS) at screening: 0-5.5, inclusive
* Neurologic stability for >/= 30 days prior to screening, and between screening and baseline
* Participants naive to prior disease-modifying therapy (DMT)
* Participants who have had at least 6 contiguous months of DMT within the past 1 year must have evidence of disease activity occurring after the full 6-month course of treatment, that is, at least one relapse or >/= 1 Gd-enhancing lesion(s) on a T1-weighted brain MRI

Exclusion Criteria:

* Known presence or suspicion of other neurologic disorders that may mimic MS, including, but not limited to, acute disseminated encephalomyelitis, neuromyelitis optica or neuromyelitis optica spectrum disorders and any neurologic, somatic, or metabolic condition that could interfere with brain function or normal cognitive or neurological development
* Patients that are aquaporin 4 positive and myelin oligodendrocyte glycoprotein (MOG) antibody positive are not eligible to participate in the study.
* In case of an ADEM-like appearance of the first MS attack, a second attack with clear MS-like features is required.
* Infection requiring hospitalization or treatment with IV anti-infective agents
* History or known presence of recurrent or chronic infection (e.g., HIV, syphilis, tuberculosis)
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to treatment allocation
* History or laboratory evidence of coagulation disorders
* Peripheral venous access that precludes IV administration and venous blood sampling
* Inability to complete a magnetic resonance imaging (MRI) scan
* History of cancer, including solid tumors, hematologic malignancies, and carcinoma in situ
* History of a severe allergic or anaphylactic reaction to humanized or murine monoclonal antibody (mAbs) or known hypersensitivity to any component of ocrelizumab solution
* Previous treatment with B-cell-targeted therapies
* Percentage of CD4 < 30%
* Absolute Neutrophil Count < 1.5x1000/microliter
* Lymphocyte count below the lower limit of normal (LLN) for age- and sex-specific reference range

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2029-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (5):
  - University of Colorado Denver Childrens Hospital Rocky Mountain MS Center, Aurora, Colorado
  - Childrens National Health Center, Washington D.C., District of Columbia
  - Boston Childrens Hospital, Boston, Massachusetts
  - Washington Universtiy school of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
- Italy (3):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - AOU Policlinico V. Emanuele - P.O G. Rodolico, Catania, Sicily
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Dzieci?cy Szpital Kliniczny im. Józefa Polikarpa Brudzi?skiego, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Mar S, Valeriani M, Steinborn B, Schreiner T, Waubant E, Filippi M, Kotulska K, Mazurkiewicz-Beldzinska M, El Azzouzi B, Lin CJ, Shen YA, Kletzl H, Evershed J, Hogea A, Manlius C, Bonati U, Banwell B. Ocrelizumab dose selection for treatment of pediatric relapsing-remitting multiple sclerosis: results of the OPERETTA I study. J Neurol. 2025 Jan 15;272(2):137. doi: 10.1007/s00415-024-12879-z. PMID 39812825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 12 investigative sites in 3 countries (the United States, Poland, and Italy). This study is still ongoing.
Pre-assignment Details: A total of 23 participants with relapsing-remitting multiple sclerosis (RRMS) received ocrelizumab per a weight-based dosing regimen.
Groups:
- Ocrelizumab 300 mg: Participants who weighed between 25 kilograms (kg) to 40 kg were administered first dose of 300 milligrams (mg) ocrelizumab as two intravenous (IV) infusions given 14 days apart i. e. 2 x 150 mg on Days 1 and 15. Participants who completed the 24-week dose exploration period were eligible to continue ocrelizumab treatment in 264-week optional ocrelizumab extension (OOE) period. Ocrelizumab 300 mg was administered as a single IV infusion given 24 weeks apart.
- Ocrelizumab 600 mg: Participants who weighed 40 kg or more were administered first dose of 600 mg ocrelizumab as two IV infusions given 14 days apart i. e. 2 x 300 mg on Days 1 and 15. Participants who completed the 24-week dose exploration period were eligible to continue ocrelizumab treatment in 264-week OOE period. Ocrelizumab 600 mg was administered as a single IV infusion given 24 weeks apart.
Period: Dose Exploration Period: 24 Week
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0
Period: OOE Period: 264 Week
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Started | 6 (Participants who completed the dose exploration period were given the option to enroll in the OOE period to receive ocrelizumab.) | 17 (Participants who completed the dose exploration period were given the option to enroll in the OOE period to receive ocrelizumab.)
Completed | 0 | 0
Not Completed | 6 | 17
Not completed — Ongoing in Study | 5 | 17
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety evaluable population included all participants who received at least one dose of study drug.
Groups:
- Ocrelizumab 300 mg: Participants who weighed between 25 kg to 40 kg were administered first dose of 300 mg ocrelizumab as two IV infusions given 14 days apart i. e. 2 x 150 mg on Days 1 and 15. Participants who completed the 24-week dose exploration period were eligible to continue ocrelizumab treatment in 264-week OOE period. Ocrelizumab 300 mg was administered as a single IV infusion given 24 weeks apart.
- Total: Total of all reporting groups
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg | Total
Number analyzed (Participants) | 6 | 17 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (0.8) | 15.3 (1.8) | 14.2 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 1 | 7 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 6 | 14 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 16 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Cluster of Differentiation (CD) 19+B cells [Median (Full Range); unit: cells/microliters (cells/µL)] — Population: Number analyzed is the number of participants with data available for analysis.
  cells/microliters (cells/µL)
    number analyzed (Participants) | 5 | 17 | 22
    (all) | 287 [160.0 to 635.0] | 234 [73.0 to 512.0] | 246 [73.0 to 635.0]

OUTCOME MEASURES:

1. Primary Outcome: Dose Exploration Period: Area Under the Concentration Versus Time Curve of Ocrelizumab
Description: The population PK model was used to simulate concentration-time course and predict individual area under the concentration versus time curve. The data for the PK parameter: area under the concentration versus time curve was collected and analyzed as per body weight range (<40kg to ≥40 kg).
Time Frame: Pre-dose 5- 30 minutes and post-dose 30 mins on Days 1, 15 and 169; At any time on Days 29, 57, 85 and 113
Population: Pharmacokinetic (PK) evaluable population included all participants who were enrolled in the study.
Measure: Median (Full Range); unit: microgram/milliters*day (µg/mL*day)
Groups:
- Body Weight < 40 kg: Participants who weighed < 40 kg were administered first dose of 300 mg ocrelizumab as two IV infusions given 14 days apart i. e. 2 x 150 mg on Days 1 and 15.
- Body Weight ≥ 40 kg: Participants who weighed ≥ 40 kg were administered first dose of 600 mg ocrelizumab as two IV infusions given 14 days apart i. e. 2 x 300 mg on Days 1 and 15.
Arm/Group | Body Weight < 40 kg | Body Weight ≥ 40 kg
Number analyzed (Participants) | 6 | 17
microgram/milliters*day (µg/mL*day) | 2187 [1565 to 3090] | 3197 [1781 to 4339]

2. Primary Outcome: Dose Exploration Period: Maximum Concentration (Cmax) of Ocrelizumab
Description: The population PK model was used to simulate concentration-time course and predict individual Cmax. The data for the PK parameter: Cmax was collected and analyzed as per body weight range (<40kg to ≥40 kg).
Time Frame: Pre-dose 5- 30 minutes and post-dose 30 mins on Days 1, 15 and 169; At any time on Days 29, 57, 85 and 113
Population: PK evaluable population included all participants who were enrolled in the study.
Measure: Median (Full Range); unit: microgram/milliters (µg/mL)
Arm/Group | Body Weight < 40 kg | Body Weight ≥ 40 kg
Number analyzed (Participants) | 6 | 17
microgram/milliters (µg/mL) | 106 [81 to 142] | 158 [113 to 209]

3. Primary Outcome: Dose Exploration Period: Levels of CD 19+ B-cell Count in Blood
Time Frame: At Week 24
Population: Safety evaluable population included all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: cells/µL
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 6 | 17
cells/µL | 91.00 [24.0 to 404.0] | 9.00 [1.0 to 151.0]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product.
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2030-12

5. Secondary Outcome: Dose Exploration Period: Level of Circulating T Cells and Natural Killer (NK) Cells
Time Frame: At Week 24
Population: Safety evaluable population included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: cells/microliter (µL)
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 6 | 17
cells/microliter (µL)
  CD3+ Total T cell | 1637.67 (578.50) | 1506.0 (468.68)
  CD4+ Helper T cell | 1044.0 (329.0) | 889.18 (252.58)
  CD8+ Cytotoxic T cell | 441.83 (180.32) | 532.65 (218.52)
  NK cells | 266.5 (182.97) | 237.76 (118.63)

6. Secondary Outcome: OOE Period: Level of Circulating T Cells and NK Cells
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2030-12

7. Secondary Outcome: Dose Exploration Period: Level of Circulating Lymphocyte, Neutrophil, Monocyte and Leukocyte
Time Frame: At Week 24
Population: Safety evaluable population included all participants who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 5 | 13
10^9 cells/L
  Lymphocyte | 1.792 (0.660) | 1.668 (0.507)
  Neutrophil | 2.60 (0.567) | 2.857 (0.762)
  Monocyte | 0.328 (0.151) | 0.343 (0.114)
  Leukocyte | 4.87 (1.35) | 5.05 (1.06)

8. Secondary Outcome: OOE Period: Level of Circulating Lymphocyte, Neutrophil, Monocyte and Leukocyte
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2030-12

9. Secondary Outcome: Developmental Milestones - Growth Velocity: Change in Height
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2030-12

10. Secondary Outcome: Developmental Milestones: Bone Age Assessment by Wrist/Hand Radiographs
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2030-12

11. Secondary Outcome: Developmental Milestones: Male and Female Puberty Assessed by Tanner Staging
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2030-12

12. Secondary Outcome: Developmental Milestones: Age at Menarche, Related With the Female Reproductive Status
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2030-12

13. Secondary Outcome: Dose Exploration Period: Number of Participants With Shift From Baseline in Non-MS Central Nervous System (CNS) Pathology as Measured by Brain Magnetic Resonance Imaging (MRI)
Description: The change in the non-MS CNS pathology was assessed using MRI scans.
Time Frame: Up to Week 24
Population: Safety evaluable population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 6 | 17
Participants | 0 | 0

14. Secondary Outcome: OOE Period: Number of Participants With Shift From Baseline in Non-MS CNS Pathology as Measured by Brain MRI
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2030-12

15. Secondary Outcome: Dose Exploration Period: Levels of Blood Immunoglobulins
Time Frame: At Week 24
Population: Safety evaluable population included all participants who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: gram/liter (g/L)
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 4 | 14
gram/liter (g/L)
  Total Immunoglobulin | 11.23 (1.40) | 11.86 (2.92)
  Immunoglobulin A | 1.27 (0.48) | 1.52 (0.61)
  Immunoglobulin G | 9.25 (1.20) | 9.73 (2.51)
  Immunoglobulin M | 0.72 (0.26) | 0.61 (0.31)

16. Secondary Outcome: OOE Period: Levels of Blood Immunoglobulins
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2030-12

17. Secondary Outcome: Dose Exploration Period: Number of Participants With Antibody Titers Against Standard Vaccines
Description: Measurement of antibody titers to common antigens (mumps, rubella, varicella, and Streptococcus pneumoniae [S. pneumoniae]) were performed.
Time Frame: At Week 24
Population: Safety evaluable population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 6 | 17
Participants
  Mumps | 0 | 0
  Pneumococcal Capsular Polysaccharides | 6 | 17
  Rubella | 0 | 0
  Varicella-Zoster Virus | 0 | 0

18. Secondary Outcome: OOE Period: Number of Participants With Antibody Titers Against Standard Vaccines
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2030-12

19. Secondary Outcome: Dose Exploration Period: Number of Participants With Anti-Drug Antibodies (ADAs) to Ocrelizumab
Time Frame: At Week 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
Number analyzed (Participants) | 6 | 17
Participants | 0 | 0

20. Secondary Outcome: OOE Period: Number of Participants With ADAs to Ocrelizumab
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2030-12

ADVERSE EVENTS:
Time Frame: Up to 3.7 years
Description: Safety population included all participants who received at least one dose of study drug. Data collected up to the primary completion date is reported here. Adverse events section will be updated one year after the study completion date.
Arm/Group | Ocrelizumab 300 mg | Ocrelizumab 600 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/17
Other Adverse Events (participants affected / at risk) | 5/6 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab 300 mg (N=6) | Ocrelizumab 600 mg (N=17)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (2)
Gonococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab 300 mg (N=6) | Ocrelizumab 600 mg (N=17)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (5) | 6 (7)
Temperature intolerance (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (4)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 11 (11)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 2 (2)
Herpes virus infection (Infections and infestations) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 7 (11)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 2 (3)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4)
Viral infection (Infections and infestations) | 0 (0) | 3 (4)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (5) | 14 (45)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Product preparation error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Torus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 1 (1)
Blood immunoglobulin M decreased (Investigations) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
CD8 lymphocytes decreased (Investigations) | 0 (0) | 1 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Fungal test positive (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 2 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Monocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain fog (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Decreased vibratory sense (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (4) | 4 (5)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (12) | 8 (29)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (2) | 3 (5)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (3) | 4 (4)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 2 (3)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT04075266/Prot_SAP_000.pdf